CLINICAL TRIAL: NCT03235817
Title: A Comparison of Different Ventilation Strategies in Infants Using the Proseal™ Laryngeal Mask Airway
Brief Title: A Comparison of Different Ventilation Strategies in Infants Using the PLMA™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00011814
Record Dates: First submitted 2013-02-08; First posted 2017-08-01 (Actual); Results first posted 2018-01-16 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2018-04

CONDITIONS: Ventilation
Keywords: Proseal™ LMA; infants; ventilation; general anesthesia; outpatient surgery
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Spontaneous ventilation (Experimental)
  Interventions: Other: Spontaneous ventilation
- Pressure support ventilation (Experimental)
  Interventions: Device: Pressure support ventilation
- Pressure control ventilation (Active Comparator)
  Interventions: Device: Pressure control ventilation

INTERVENTIONS:
Other: Spontaneous ventilation — The patient will breathe spontaneously (on their own) while under general anesthesia throughout the duration of the surgery.
  Arms: Spontaneous ventilation
Device: Pressure support ventilation — The patient will breathe on their own and with a little assistance from the anesthesia machine while under general anesthesia throughout the duration of the surgery.
  Arms: Pressure support ventilation
Device: Pressure control ventilation — The patient's ventilation will be completely supported by the anesthesia machine while under general anesthesia throughout the duration of the surgery.
  Arms: Pressure control ventilation

SUMMARY:
The purpose of this research study is to compare difference between breathing by oneself or with the partial help from an anesthesia machine in infants under general anesthesia.

Hypothesis: Infants undergoing general anesthesia with a PLMA™ will be better ventilated (improved breathing) with the help of the breathing machine versus breathing on their own.

DETAILED DESCRIPTION:
The laryngeal mask airway (LMA) is a breathing device that sits above the vocal cords and allows the patient to breathe in and out adequately under general anesthesia (GA). The ProSeal™ laryngeal mask airway (PLMA™) is a specialized type of LMA with a design that permits the delivery of higher pressures to help the patient breathe in and out (ventilate) and also contains a channel to suction the stomach.

Infants under GA may breathe through a PLMA in different ways. Spontaneous ventilation consists of the infants breathing on their own through a PLMA™. Pressure support ventilation allows the patient to breathe on their own with additional help from the anesthesia machine. Pressure control ventilation allows the patient to breathe with the help of an anesthesia machine.

An infant undergoing surgery requires a deep level of general anesthesia which negatively affects their ability to ventilate. Thus, infants may not breathe in oxygen and carbon dioxide out adequately at this level of anesthesia and it may be beneficial to provide some level of support to enhance carbon dioxide exchange and to avoid hypoventilation.

This study will attempt to determine whether pressure support ventilation improves ventilation in infants undergoing outpatient surgery.

ELIGIBILITY:
Inclusion Criteria:

1. ASA (American Society of Anesthesiologists) physical classification of 1 or 2
2. Outpatient surgical procedures
3. Surgical procedure anticipated to be < 90 minutes
4. Subject age of 1 - 11 months (inclusive)

Exclusion Criteria:

1. Inpatient- Such individuals may have underlying disease processes which puts them at an increased risk under general anesthesia for hypoventilation
2. ASA physical classification of 3, 4 or E
3. Premature infants or infants < 44 weeks post-conceptual age
4. Risk of aspiration- Intubation with an endotracheal tube may be required for general anesthesia.
5. Patients with malignant hyperthermia or family history of malignant hyperthermia- Administration of inhalational agents for general anesthesia is contraindicated.
6. Patients with tracheostomies- The individual's airway is already established and PLMA™ placement is not required.

Ages: 1 Month to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2009-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Templeton, M.D., Principal Investigator — Wake Forest
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Brain AI, McGhee TD, McAteer EJ, Thomas A, Abu-Saad MA, Bushman JA. The laryngeal mask airway. Development and preliminary trials of a new type of airway. Anaesthesia. 1985 Apr;40(4):356-61. PMID 4003736

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Spontaneous Ventilation | Pressure Support Ventilation | Pressure Control Ventilation
Started | 13 | 13 | 13
Completed | 10 | 12 | 11
Not Completed | 3 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spontaneous Ventilation | Pressure Support Ventilation | Pressure Control Ventilation | Total
Number analyzed (Participants) | 10 | 12 | 11 | 33
Age, Customized [Mean (Standard Deviation); unit: months]
  Age | 7.1 (2) | 7.3 (2) | 6.9 (1.9) | 7.1 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 3
  Male | 10 | 11 | 9 | 30
Weight [Mean (Standard Deviation); unit: kg] | 8 (1.7) | 8.5 (.9) | 8.2 (1.3) | 8.2 (1.4)
PLMA Size (ProSeal laryngeal mask airway) [Count of Participants; unit: Participants]
  Size 1.5 | 8 | 10 | 8 | 26
  Size 2 | 2 | 2 | 3 | 7
Induction Time [Mean (Standard Deviation); unit: minutes] | 9.5 (5.9) | 8.6 (3.3) | 9.6 (3.1) | 9.2 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Mean Values of End-tidal Carbon Dioxide and Tidal Volume Compared Between the Spontaneous Ventilation and Pressure Support Ventilation Groups.
Description: Mean values of end-tidal carbon dioxide (ETCO2) and tidal volume (TV) between 5 and 45 minutes compared between the spontaneous ventilation (SV) and pressure support ventilation groups (PSV).
Time Frame: Up to 45 minutes
Measure: Mean (Standard Deviation); unit: cc/kg
Arm/Group | Spontaneous Ventilation | Pressure Support Ventilation
Number analyzed (Participants) | 10 | 12
cc/kg
  Mean Values of Tidal Volume | 4.5 (.3) | 7 (.5)
  Mean Values of End-Tidal Carbon Dioxide | 51.8 (2.9) | 49 (1.5)

2. Primary Outcome: Mean Values of ETCO2 and TV Compared Between the SV and PCV Groups
Description: Mean values of ETCO2 and TV between 5 and 45 minutes compared between the SV and Pressure control ventilation (PCV) groups.
Time Frame: Up to 45 minutes
Measure: Mean (Standard Deviation); unit: cc/kg
Arm/Group | Spontaneous Ventilation | Pressure Control Ventilation
Number analyzed (Participants) | 10 | 11
cc/kg
  ETCO2 | 51.8 (2.9) | 48.3 (1.6)
  TV | 4.5 (0.3) | 7.0 (0.4)

3. Primary Outcome: Mean Values of ETCO2 and TV Compared Between the PSV and PCV Groups
Description: Mean values of ETCO2 and TV between 5 and 45 minutes compared between the PSV and PCV groups
Time Frame: up to 45 minutes
Measure: Mean (Standard Deviation); unit: cc/kg
Arm/Group | Pressure Support Ventilation | Pressure Control Ventilation
Number analyzed (Participants) | 12 | 11
cc/kg
  ETCO2 | 49.0 (1.5) | 48.3 (1.6)
  TV | 7.0 (0.5) | 7.0 (0.4)

4. Secondary Outcome: Mean Values of Respiratory Rates Between Spontaneous Ventilation and Pressure Support Ventilation Groups.
Description: Mean values of respiratory rate between 5 and 45 minutes compared between spontaneous ventilation and pressure support ventilation groups.
Time Frame: Up to 45 minutes
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Spontaneous Ventilation | Pressure Support Ventilation
Number analyzed (Participants) | 10 | 12
breaths per minute | 32.2 (2.2) | 25.1 (.8)

5. Secondary Outcome: Mean Values of Respiratory Rate Compared Between the Spontaneous Ventilation and Pressure Control Ventilation Groups.
Description: Mean values of respiratory rate between 5 and 45 minutes compared between the spontaneous ventilation and pressure control ventilation groups.
Time Frame: Up to 45 minutes
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Spontaneous Ventilation | Pressure Control Ventilation
Number analyzed (Participants) | 10 | 11
breaths per minute | 32.2 (2.2) | 22.3 (1.2)

6. Secondary Outcome: Mean Values of Respiratory Rate Compared Between Pressure Support Ventilation and Pressure Control Ventilation Groups.
Description: Mean values of respiratory rate between 5 and 45 minutes compared between pressure support ventilation and pressure control ventilation groups.
Time Frame: Up to 45 minutes
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Pressure Support Ventilation | Pressure Control Ventilation
Number analyzed (Participants) | 12 | 11
breaths per minute | 25.1 (.8) | 22.3 (1.2)

ADVERSE EVENTS:
Arm/Group | Spontaneous Ventilation | Pressure Support Ventilation | Pressure Control Ventilation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes